CLINICAL TRIAL: NCT06572124
Title: Clinical Performance of Universal Adhesive with and Without Acid Resistant Silane Coupling Agent in Carious Cervical Lesions :A Randomized Controlled Trial
Brief Title: Clinical Performance of ARS Containing Universal Adhesives in Carious Cervical Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed El-Kotaby, Prinicipal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU ARS
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Carious Lesion; Cervical Caries
MeSH Terms: conditions — Dental Caries; Root Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Universal adhesive without acid resistant silane coupling agent (Active Comparator): Universal adhesive with normal silane (comparator) After the acid etching and rinsing and drying step, the universal adhesive with normal silane will be actively applied for 20 second , then light cured for 20 seconds then the restoration will be placed
  Interventions: Procedure: universal adhesive without Acid resistant silane coupling agent
- Universal adhesive with acid resistant silane coupling agent (Experimental): Universal adhesive with acid resistant silane coupling agent (Intervention) After the acid etching and rinsing and drying step, the universal adhesive with acid resistant silane coupling agent will be actively applied for 20 second , then light cured for 20 seconds then the restoration will be placed
  Interventions: Procedure: universal adhesive with Acid resistant silane coupling agent

INTERVENTIONS:
Procedure: universal adhesive without Acid resistant silane coupling agent — After cavity preparations, enamel margins will be etched for 30 seconds then rinsed and dried, then the Universal adhesive without acid resistant silane coupling agent will be actively applied for 20 seconds then air thinned for 5 seconds then cured for 20 seconds.Then the composite restoration will be placed.
  Arms: Universal adhesive without acid resistant silane coupling agent
Procedure: universal adhesive with Acid resistant silane coupling agent — After cavity preparations, enamel margins will be etched for 30 seconds then rinsed and dried, then the Universal adhesive which contains acid resistant silane coupling agent will be actively applied for 20 seconds then air thinned for 5 seconds then cured for 20 seconds.Then the composite restoration will be placed.
  Arms: Universal adhesive with acid resistant silane coupling agent

SUMMARY:
Evaluation of composite restorations done in carious cervical lesions restored by a conventional universal adhesive in comparison to a universal adhesive that contains and resistant silane coupling agent according to the Modified United States Public Health Service (USPHS) criteria over 18 months.

DETAILED DESCRIPTION:
The presence of acidic monomers in the bottle during storage can lead to the hydrolysis of silane contained in universal adhesives, potentially reducing its effectiveness and causing instability,The acid resistant silane coupling agent has a protective structure against attacks from acidic monomers. Therefore, long-term storage stability can be expected by suppressing hydrolysis. The protective structure is removed when the concentration of acidic monomers increases by air drying after application. This activates ARS, exerting the silane coupling effect.

ELIGIBILITY:
Inclusion Criteria:

* Participants Inclusion:

  • Adults aging from 21-67 years old who were in need of restoration of at least one notch-shaped cervical lesion
* Teeth Inclusion:

  * Vital teeth with carious cervical lesions in incisors , canines ,premolars& molars

Exclusion Criteria:

* Participants Exclusion:

  * Patients with fewer than 20 teeth
  * Poor oral hygiene
  * Uncontrolled periodontal disease
  * Xerostomia
  * Known allergy to resin-based materials
  * Medically compromised, pregnant, or breast-feeding
* Teeth Exclusion:

  * Non vital teeth
  * Teeth that are out of occlusion
  * Previously restored teeth

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Retention (Success rate) | T0=baseline 24 hours postoperative. T1=12 months postoperative. T2=18 months postoperative.
  Alpha (A) Present Bravo (B) Partial loss but clinically acceptable Charlie (C)Clinically unacceptable partial loss or absent

SECONDARY OUTCOMES:
Marginal adaptation | T0=baseline 24 hours postoperative. T1=12 months postoperative. T2=18 months postoperative.
  Alpha (A) Restoration adapts closely to the tooth structure; there is no visible crevice.
  Bravo (B) There is a visible crevice, the explorer will penetrate, without dentin exposure.
  Charlie(C)The explorer penetrates into a crevice in which dentin or the base is exposed.
Marginal discoloration | T0=baseline 24 hours postoperative. T1=12 months postoperative. T2=18 months postoperative.
  Alpha (A) No marginal discoloration. Bravo (B) Minor marginal discoloration without staining toward the pulp, only visible using a mirror and operating light.
  Charlie(C) Deep discoloration with staining toward the pulp, visible at a speaking distance of 60 to 100 cm.
Secondary caries | T0=baseline 24 hours postoperative. T1=12 months postoperative. T2=18 months postoperative.
  Alpha (A) No active caries present Charlie(C) Active caries is present in contact with the restoration

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No